CLINICAL TRIAL: NCT04154098
Title: Evaluation of a Method to Support Unstable Shoulders by Means of a Textile Scapula Orthosis
Brief Title: Evaluation of a Textile Scapula Orthosis
Acronym: ScapOrthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ScapulaOrthosis_v1
Record Dates: First submitted 2019-10-23; First posted 2019-11-06 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Muscular Dystrophies; Scapular Dyskinesis; Muscular Dystrophy, Facioscapulohumeral; Muscle Weakness; Muscular Weakness; Muscular Dystrophy
Keywords: Scapula alata; Scapular winging; Scapula orthosis; Range of Motion; Movement control; Manual Scapula Assistance
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Facioscapulohumeral; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: All patients perform the experiment in all conditions. The without orthosis, with orthosis and manual assistance conditions will be presented in randomized order, followed by the functional task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- NO-OA-MA-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test
- NO-MA-OA-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test
- OA-NO-MA-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test
- OA-MA-NO-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test
- MA-NO-OA-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test
- MA-OA-NO-FT (Experimental): Participants elevate their arm without assistance (NO) - with orthosis assistance (OA) - with manual assistance (MA) in the given order, followed by the functional task (FT)
  Interventions: Device: Scapula orthosis assistance; Procedure: Manual scapula assistance; Other: No assistance; Other: Functional Test

INTERVENTIONS:
Device: Scapula orthosis assistance — Participants are elevating their arm while their scapula is assisted by the scapula orthosis
  Other Names: OA
Procedure: Manual scapula assistance — Participants are elevating their arm while their scapula is assisted by a trained personnel
  Other Names: MA
Other: No assistance — Participants are elevating their arm without being assisted
Other: Functional Test — Participants perform a functional test once without (NO) and once with (OA) the orthosis
  Other Names: FT

SUMMARY:
Shoulder instability due to muscle weakness is a common problem in disorders of the upper extremities. During arm motion, the scapula acts as a dynamic base for the humeral head. To safely move the shoulder with an exoskeleton for the upper extremities a textile orthosis was developed that stabilizes the scapula against the thorax. The support level of the orthosis is continuously manually adjustable. To test the feasibility of our design and to improve the functionality of the textile orthosis, it needs to be investigated how the orthosis acts on people affected by shoulder instability. The investigators seek to explore how people with shoulder instability respond to the orthosis, and how they may benefit from the orthosis function. Therefore, the range of motion of arm elevation will be compared in different conditions: (i) without any support, (ii) with the support of a trained therapist, and (iii) when the device is engaged at the individual's optimal support level. Additionally, pilot tests will be performed to fix different parameters in our study protocol, such as the the optimal orthosis stiffness level and the ideal number of movement repetitions.

DETAILED DESCRIPTION:
In this study, participants suffering from muscular weakness in the upper extremities, particularly the shoulder joint, will be recruited. A clear indicator for muscular weakness in the shoulder joint is a scapula alata (winging scapula). Hence, participants recruited for this study should present with a scapula alata and a limited RoM of at least one of their upper extremities.

This study is designed as a cross-over trial. Each participant will take part in an experimental session that will last approximately 2 hours. At the beginning of the experiment, the participant will be informed about the measurement and sign the informed consent sheet. Additional demographic data and level of ability will be collected in a questionnaire.

Before the measurements, participants will be fitted a textile scapula orthosis. The orthosis will be instrumented to quantify the amount of support the orthosis provides to the user. Therefore, an array of force sensors is mounted between the orthosis and the skin to measure the qualitative force distribution and its rate of change. To measure the absolute force applied to the plate, a load cell will be mounted on the orthosis fastening mechanism. All force data will be collected synchronously through a Micro-Controller board.

The participants will be equipped with reflective adhesive markers to define the reference points for the range of motion measurements, which will be done with a goniometer and photographic opto-electronic motion tracking.

Nine blocks of measurements will be conducted, lasting 5 minutes each. The remaining time in the study accounts for rest periods, the mounting and demounting of the orthosis, instructions and questionnaires. The first eight blocks will present the following treatment conditions in randomized order:

* No support (NO): the scapula is not assisted during arm elevation.
* Manual scapular assistance (SA): a trained person assists the scapula during arm elevation manually.
* Orthosis support (OS): the scapula is assisted by the textile orthosis set to meaningfully different force levels.
* Motor control task (MT): The participant reaches for a target placed at the maximum elevation height in the NO condition, once without and once with the orthosis.

While one block each is performed in the NO, SA and MT conditions, six blocks are performed in the OS condition with the orthosis set to meaningfully different force levels.

In each measurement set, participants will elevate their arms in one of two planes of horizontal rotation:

* 30° (R30) as measured from the coronal body plane.
* 80° (R80) as measured from the coronal body plane.

During arm elevation, the arm is fully extended, i.e. the elbow and wrist are fully stretched. In this position, the center of mass has the largest lever arm and therefore the maximum torque due to gravity occurs in the shoulder. One measurement set will be done in each elevation plane. During the OS condition, the orthosis will be opened between measurement sets to allow for comfort and unhindered breathing and to guarantee independence of measurement data.

After the experiment, the perceived exertion and orthosis comfort will be assessed using the Borg Scale and the Nordic Questionnaire.

Before the study, several study parameters will be determined in pilot studies with variable duration, not exceeding 2 hours. The participants in the pilot studies and the final study might be identical. During the pilot tests, participants will wear an orthosis similar to the one used in the study. Hence, effort and strain for participants will be equal or less to the final study. The pilot tests include

* Definition of optimal pressure and protocol to consistently find this pressure.
* Definition of optimal orthosis configuration.
* Definition of repeatability when orthosis is unmounted and mounted again.
* Definition of meaningful difference between pressure levels.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed scapula alata (winging scapula)
* Limited range of motion of at least one of the upper extremities.
* Ability to elevate the arm at least 110° passively
* Able to sit in a chair without additional support and without leaning on the back rest.

Exclusion Criteria

* Frozen shoulder
* Osteoporosis or arthrosis of the shoulder joint
* Shoulder subluxation
* Excessive spasticity of the affected arm
* Skin ulcerations on the paretic arm or torso
* Known risk for impingement
* Orthopaedic, rheumatological or other disease restricting movements of the paretic arm
* Pain or stiffness in the shoulder joint limiting their movement
* Cardiopulmonary disease
* Psychiatric disorders or severe cognitive impairments that limit their ability to understand the study instructions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Range of motion of arm elevation | Up to 2 hours per participant
  The maximum angle of arm elevation in the 80 or 30 degree plane the participant can reach under the different study conditions
Improvement of range of motion of arm elevation | Up to 2 hours per participant
  The relative or absolute improvement of arm elevation in the orthosis assistance condition when compared to the without assistance condition and/or the manual assistance condition
Range of motion of arm elevation for different force levels in the orthosis assistance condition | Up to 2 hours per participant
  Relative or absolute improvement in range of motion or range of motion of arm elevation for different force levels in the orthosis assistance condition
Motor control during functional task | Up to 2 hours per participant
  Assessment of kinematic variables such as movement smoothness during the functional task

SECONDARY OUTCOMES:
Beneficiary or Responsiveness level | Up to 2 hours per participant
  Identification of beneficiary/responsiveness threshold in the correlation between range of motion of arm elevation with orthosis assistance and without assistance
Threshold for Beneficiary or Responsiveness level | Up to 2 hours per participant
  Correlation between beneficiary/responsiveness level and level of disability as assessed by the Manual Muscle Test (MMT, Jepsen 2004) and/or the Range of Motion Test (Nadeau 2007)
Perceived effort | Up to 2 hours per participant
  Perceived effort (Borg Scale) of arm elevation for the different study conditions
Motor control during arm elevation | Up to 2 hours per participant
  Assessment of kinematic variables such as movement smoothness for the different study conditions
Comfort | Up to 2 hours per participant
  Assessment and comparison of discomfort during the different conditions (Modified short version of the Nordic Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof., Principal Investigator — ETH Zurich
Locations (2):
- Kliniken Schmieder Konstanz, Konstanz, Basen-Wuerttemberg, Germany
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veeger HE, van der Helm FC. Shoulder function: the perfect compromise between mobility and stability. J Biomech. 2007;40(10):2119-29. doi: 10.1016/j.jbiomech.2006.10.016. Epub 2007 Jan 12. PMID 17222853
- [Background] Paine RM, Voight M. The role of the scapula. J Orthop Sports Phys Ther. 1993 Jul;18(1):386-91. doi: 10.2519/jospt.1993.18.1.386. PMID 8348140
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] Orrell RW, Copeland S, Rose MR. Scapular fixation in muscular dystrophy. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD003278. doi: 10.1002/14651858.CD003278.pub2. PMID 20091543
- [Background] Vastamaki M, Pikkarainen V, Vastamaki H, Ristolainen L. Scapular Bracing is Effective in Some Patients but Symptoms Persist in Many Despite Bracing. Clin Orthop Relat Res. 2015 Aug;473(8):2650-7. doi: 10.1007/s11999-015-4310-1. Epub 2015 Apr 25. PMID 25910775
- [Background] Barnett ND, Mander M, Peacock JC, Bushby K, Gardner-Medwin D, Johnson GR. Winging of the scapula: the underlying biomechanics and an orthotic solution. Proc Inst Mech Eng H. 1995;209(4):215-23. doi: 10.1243/PIME_PROC_1995_209_348_02. PMID 8907215
- [Background] Jepsen J, Laursen L, Larsen A, Hagert CG. Manual strength testing in 14 upper limb muscles: a study of inter-rater reliability. Acta Orthop Scand. 2004 Aug;75(4):442-8. doi: 10.1080/00016470410001222-1. PMID 15370589
- [Background] Nadeau S, Kovacs S, Gravel D, Piotte F, Moffet H, Gagnon D, Hebert LJ. Active movement measurements of the shoulder girdle in healthy subjects with goniometer and tape measure techniques: a study on reliability and validity. Physiother Theory Pract. 2007 May-Jun;23(3):179-87. doi: 10.1080/09593980701209246. PMID 17558881
- [Derived] Georgarakis AM, Xiloyannis M, Dettmers C, Joebges M, Wolf P, Riener R. Reaching higher: External scapula assistance can improve upper limb function in humans with irreversible scapula alata. J Neuroeng Rehabil. 2021 Sep 3;18(1):131. doi: 10.1186/s12984-021-00926-z. PMID 34479574